CLINICAL TRIAL: NCT03315715
Title: Dynamic Magnetic Resonance Imaging Following Vaginal Reconstructive Surgery; a Prospective Study to Describe Anatomy
Brief Title: Dynamic Magnetic Resonance Imaging Before and After Vaginal Prolapse Repair
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 17-061
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2019-11

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to describe the impact of vaginal reconstruction, including an intraperitoneal vaginal vault suspension for pelvic organ prolapse (POP) on pelvic anatomy using dynamic magnetic resonance imaging (MRI) of the pelvis.

DETAILED DESCRIPTION:
Approximately 1 in 11 women will undergo surgery for POP by age 80 years. POP occurs due to a defect or weakness of the pelvic floor, resulting in the herniation of pelvic organs through the vagina. The goal of surgical interventions has historically been thought to restore normal pelvic anatomy. Restoration of pelvic anatomy has been demonstrated following pelvic reconstructive surgery by way of significantly improved postoperative Pelvic Organ Prolapse Quantification (POPQ) scale measurements. Furthermore, improved POPQ measurements have also been shown to be positively correlated with improved patient satisfaction.

More recently, attention has turned toward using imaging studies to describe the postoperative anatomical changes seen in pelvic reconstructive surgery. The purpose of this study is to describe the impact of vaginal reconstruction, including an intraperitoneal vaginal vault suspension for POP on pelvic anatomy using dynamic MRI of the pelvis.

The primary aim is to compare postoperative dynamic pelvic MRI measurements to preoperative measurements in patients who undergo prolapse repair vaginally including anterior, posterior and intraperitoneal vaginal vault suspension repairs for POP.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* English-speaking
* Undergoing anterior, posterior and intraperitoneal vaginal vault suspension by a physician at Cincinnati Urogynecology Associates, TriHealth for the treatment of symptomatic POP
* Concomitant procedures such as hysterectomy, suburethral sling, bilateral salpingectomy or salpingooophorectomy
* Willingness to participate in study

Exclusion Criteria:

* Unwillingness to participate in the study
* Pregnancy
* Contraindication to pelvic MRI, such as a metal implanted device (excluding titanium) or claustrophobia
* Previous surgery for apical prolapse such as sacrocolpopexy or vaginal vault suspension, or transvaginal mesh for prolapse
* Physical or mental impairment that would affect the subject's ability to complete the dynamic MRI, including patient's with dementia or those who have impaired mobility
* Known findings that may distort pelvic anatomy, such as a pelvic mass, congenital anomaly, or history of pelvic radiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women 18 years of age or older, who undergo intraperitoneal vaginal vault suspension, with or without additional concomitant procedures by a physician at Cincinnati Urogynecology Associates, TriHealth for treatment of POP.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2020-05-24 (Actual)

PRIMARY OUTCOMES:
Change in H-line, Dynamic MRI measurement between pre- and post | Before surgery and 12 weeks after surgery
  The distance from pubic symphysis to the posterior anal canal
Change in M-line, Dynamic MRI measurement | Before surgery and 12 weeks after surgery
  The descent of the levator plate from the pubococyygeal line (PCL)
Change in O classification | Before surgery and 12 weeks after surgery
  The type of visceral prolapse (cystocele, rectocele, enterocele and the degree beyond the H-line

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- TriHealth - Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No